CLINICAL TRIAL: NCT06549309
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics of JMKX003801 in Healthy Participants
Brief Title: Trial of JMKX003801 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JMKX003801-101
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): JMKX003801
  Interventions: Drug: JMKX003801
- Placebo Comparator (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JMKX003801 — For Ascending Single Dose of JMKX003801，Five（5）cohorts of 40 participants (each cohort contains 6 active and 2 placebo) are planned for evaluation.
  For Ascending Multiple Dose of JMKX003801，Three（3）cohort of 30 participants (each cohort contains 8 active and 2 placebo) are planned for evaluation.
  Arms: Experimental
Drug: Placebo — For Ascending Single Dose of JMKX003801，Five（5）cohorts of 40 participants (each cohort contains 6 active and 2 placebo) are planned for evaluation.
  For Ascending Multiple Dose of JMKX003801，Three（3）cohorts of 30 participants (each cohort contains 8 active and 2 placebo) are planned for evaluation.
  Arms: Placebo Comparator

SUMMARY:
To Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of JMKX003801 Administered Randomly, Double-blind, Placebo-controlled, Single-ascending Dose and Multiple-ascending Dose in Chinese Healthy Adult Participants

ELIGIBILITY:
Inclusion Criteria:

* The subjects have a thorough understanding of the study content, process, and potential adverse effects, and are willing to complete the study according to the requirements of the experimental protocol;
* Healthy adult males and/or females, 18 to 45 years of age;
* Body mass index (BMI) ≥ 19 and ≤ 28.0 (kg/m2) ,weight ≥45kg (female) or ≥50kg (male) .

Exclusion Criteria:

* Had or currently have serious clinical diseases related to circulatory system, respiratory system, digestive system, nervous system, endocrine system, blood lymphatic system, genitourinary system or psychiatry, or any other diseases judged by investigators that will be interference to the results of this study;
* Use of any over-the-counter (OTC) medication, prescription medicine, Chinese herbal medicine , within 2 weeks prior to the time of informed consent signed;
* Pregnant or lactating women;
* Other conditions unsuitable for the trial judged by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From baseline to Day 3
  Incidence and features of AEs

SECONDARY OUTCOMES:
Serum concentrations of JMKX003801 | From baseline to Day 3
  Serum concentrations of JMKX003801

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No